CLINICAL TRIAL: NCT00393367
Title: Budesonide Inhalation Suspension for Acute Asthma in Children
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2006-8-4875
Record Dates: First submitted 2006-10-25; First posted 2006-10-27 (Estimated); Results first posted 2011-07-25 (Estimated); Last update posted 2012-08-10 (Estimated); Status verified 2012-08

CONDITIONS: Asthma; Acute Asthma; Reactive Airway Exacerbation
Keywords: Asthma; Acute; Treatment; Children; Pediatric; Inhaled corticosteroid; Budesonide; Budesonide inhalation suspension; Asthma score; Emergency; Emergency Department; Asthma flare; Clinical trial; Randomized clinical trial; Randomized trial; Pulmonary index score; Hospitalization; Moderate asthma; Severe asthma; Mixing budesonide; Budesonide admixture; Albuterol; Continuous albuterol; Ipratropium bromide
MeSH Terms: conditions — Asthma; Emergencies | interventions — Albuterol; Budesonide; Prednisolone; Prednisone; Methylprednisolone; Ipratropium

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Saline Placebo (Placebo Comparator): All subjects will receive 3 albuterol sulfate doses, 2 ipratropium bromide doses, and systemic corticosteroids. All patients will receive both the systemic corticosteroids and one dose of a mixture of albuterol and ipratropium bromide while guardians are approached for consent. Patients randomized to this placebo comparator arm will then receive 2 nebulized albuterol doses mixed with 8mL of normal saline. Finally, all patients will receive the second nebulized ipratropium dose.
  Interventions: Drug: Prednisolone, prednisone, or methylprednisolone; Drug: Albuterol, ipratropium bromide; Drug: Ipratropium bromide
- Budesonide Inhalaiton Suspension (Experimental): All subjects will receive 3 albuterol sulfate doses, 2 ipratropium bromide doses, and systemic corticosteroids. All patients will receive both the systemic corticosteroids and one dose of a mixture of albuterol and ipratropium bromide while guardians are approached for consent. Patients randomized to this intervention arm will then receive 2 nebulized albuterol doses mixed with 8mL of budesonide inhalation suspension (BIS). Finally, all patients will receive the second nebulized ipratropium dose.
  Interventions: Drug: Budesonide inhalation suspension (0.5 mg/2mL) 2mg, albuterol (5mg/mL) 7.5 or 10mg; Drug: Prednisolone, prednisone, or methylprednisolone; Drug: Albuterol, ipratropium bromide; Drug: Ipratropium bromide

INTERVENTIONS:
Drug: Budesonide inhalation suspension (0.5 mg/2mL) 2mg, albuterol (5mg/mL) 7.5 or 10mg — Patients randomized to budesonide inhalation suspension (BIS) receive 2 nebulized albuterol sulfate (5mg/mL) doses (2mL =10mg for patients over 20kg, 1.5mL =7.5mg for patients 10-20kg) mixed with 8mL (2mg) of BIS(0.5mg/2mL). The albuterol sulfate and BIS mixture is delivered by a medium volume, high flow nebulizer (AirLife Mister FinityTM)with an oxygen flow rate of 8L/min via a tight-fitting face mask.
  Other Names: Pulmicort; Albuterol
  Arms: Budesonide Inhalaiton Suspension
Drug: Prednisolone, prednisone, or methylprednisolone — All patients are given 2mg/kg of systemic corticosteroids (max 60mg). Patients who can tolerate pills are given oral prednisone, those who cannot are given oral prednisolone, and those who cannot tolerate oral medications are given IV methylprednisolone.
  Other Names: Prednisolone; prednisone; methylprednisolone
Drug: Albuterol, ipratropium bromide — While guardians are approached for possible participation, patients are given a single nebulized dose of albuterol sulfate (5mg/mL) mixed with ipratropium bromide (500mcg/2.5mL). Patients who weigh 10-20kg receive 3.75mg of albuterol. Patients over 20kg receive 5mg of albuterol. All patients receive 500mcg of ipratropium bromide. Albuterol sulfate and ipratropium bromide are delivered by a medium volume, high flow nebulizer (AirLife Mister FinityTM)with an oxygen flow rate of 8L/min via a tight-fitting face mask.
  Other Names: Albuterol; Atrovent
Drug: Ipratropium bromide — 500 mcg/2.5mL. All patients receive a final dose of ipratropium bromide after the intervention or placebo. The ipratropium bromide is delivered by a medium volume, high flow nebulizer (AirLife Mister FinityTM) with an oxygen flow rate of 8L/minute via a tight-fitting face mask.
  Other Names: Atrovent

SUMMARY:
The purpose of this study is to determine whether the addition of budesonide inhalation suspension (BIS) to the standard therapy of albuterol, ipratropium bromide, and systemic corticosteroids (SCS) for moderate to severe asthma flares in children reduces asthma severity more rapidly than standard therapy alone.

DETAILED DESCRIPTION:
Context: Acute asthma is a leading cause of emergency department (ED) visits and hospitalizations. Although standard therapy for acute asthma includes systemic corticosteroids (SCS), these drugs take many hours to have an effect. Recent studies demonstrate that inhaled corticosteroids (ICS) may improve patients' asthma severity more rapidly than SCS and may decrease hospitalizations. Only a few small studies have evaluated ICS added to standard therapy for acute asthma in children.

Objective: To determine if adding the nebulized steroid budesonide to standard therapy including SCS improves patients' asthma severity faster than standard therapy alone and leads to fewer hospitalizations.

Study Design/Setting/Participants: A double-blind, randomized, controlled trial of budesonide inhalation suspension (BIS) versus placebo for children 2 to 18 years of age who present to a tertiary care, urban pediatric ED with a moderate to severe asthma flare.

Intervention: Participants will receive standard therapy including SCS, albuterol, and ipratropium bromide and will be randomly assigned to also receive either nebulized BIS or saline.

Study Measures: Differences in asthma scores, vital signs, and the need for hospitalization will be compared between treatment groups.

ELIGIBILITY:
Inclusion Criteria:

* Chief complaint of "respiratory distress", "asthma", "trouble breathing", or "reactive airway disease"
* Males or females age 2 to 18 years
* Weight greater than or equal to 10 kilograms
* Two or more prior Emergency Department or primary care visits for asthma or reactive airway disease
* Identified in triage as either "acute" or "critical"
* Asthma score of 8 or greater
* Systemic corticosteroid prescribed in the Emergency Department
* English-speaking parent/guardian present
* Parental/guardian permission (informed consent) and if appropriate, child assent

Exclusion Criteria:

* Systemic corticosteroid use in the last 30 days
* Chronic lung diseases including cystic fibrosis
* Sickle cell anemia
* Immunodeficiency
* Cardiac disease requiring surgery or medications
* Adverse drug reaction or allergy to budesonide, albuterol, ipratropium bromide, prednisone, prednisolone, or methylprednisolone
* Known renal or hepatic dysfunction
* Exposure to varicella in the last 21 days
* Impending respiratory failure requiring positive pressure ventilation
* Altered level of consciousness
* Suspected foreign body aspiration or croup
* Prior enrollment in the study

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 179 (Actual)
Dates: Start 2006-12; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia J Mollen, M.D., Principal Investigator — Children's Hospital of Philadelphia; Bryan D. Upham, M.D., Study Director — University of New Mexico Children's Hospital
Locations (1):
- Children's Hospital of Philadelphia Emergency Department, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Edmonds ML, Camargo CA Jr, Pollack CV Jr, Rowe BH. Early use of inhaled corticosteroids in the emergency department treatment of acute asthma. Cochrane Database Syst Rev. 2003;(3):CD002308. doi: 10.1002/14651858.CD002308. PMID 12917930
- [Background] Qureshi F, Pestian J, Davis P, Zaritsky A. Effect of nebulized ipratropium on the hospitalization rates of children with asthma. N Engl J Med. 1998 Oct 8;339(15):1030-5. doi: 10.1056/NEJM199810083391503. PMID 9761804
- [Background] Sung L, Osmond MH, Klassen TP. Randomized, controlled trial of inhaled budesonide as an adjunct to oral prednisone in acute asthma. Acad Emerg Med. 1998 Mar;5(3):209-13. doi: 10.1111/j.1553-2712.1998.tb02614.x. PMID 9523927
- [Background] Devidayal, Singhi S, Kumar L, Jayshree M. Efficacy of nebulized budesonide compared to oral prednisolone in acute bronchial asthma. Acta Paediatr. 1999 Aug;88(8):835-40. doi: 10.1080/08035259950168748. PMID 10503681
- [Background] Scarfone RJ, Loiselle JM, Wiley JF 2nd, Decker JM, Henretig FM, Joffe MD. Nebulized dexamethasone versus oral prednisone in the emergency treatment of asthmatic children. Ann Emerg Med. 1995 Oct;26(4):480-6. doi: 10.1016/s0196-0644(95)70118-4. PMID 7574132
- [Background] Nuhoglu Y, Atas E, Nuhoglu C, Iscan M, Ozcay S. Acute effect of nebulized budesonide in asthmatic children. J Investig Allergol Clin Immunol. 2005;15(3):197-200. PMID 16261956
- [Background] Schuh S, Reisman J, Alshehri M, Dupuis A, Corey M, Arseneault R, Alothman G, Tennis O, Canny G. A comparison of inhaled fluticasone and oral prednisone for children with severe acute asthma. N Engl J Med. 2000 Sep 7;343(10):689-94. doi: 10.1056/NEJM200009073431003. PMID 10974132

RESULTS

PARTICIPANT FLOW:
Groups:
- Budesonide Inhalation Suspension (BIS): standardized treatment with nebulized Budesonide Inhalation Suspension (BIS)
- Placebo (Saline): standardized treatment with nebulized saline
Period: Overall Study
Arm/Group | Budesonide Inhalation Suspension (BIS) | Placebo (Saline)
Started | 91 | 88
Completed | 89 | 81
Not Completed | 2 | 7
Not completed — Protocol Violation | 2 | 5
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Budesonide Inhalation Suspension (BIS) | Placebo (Saline) | Total
Number analyzed (Participants) | 91 | 88 | 179
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 91 | 88 | 179
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 6.2 (3.9) | 6.3 (4.0) | 6.2 (4.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 34 | 61
  Male | 64 | 54 | 118
Region of Enrollment [Number; unit: participants]
  United States | 91 | 88 | 179

OUTCOME MEASURES:

1. Primary Outcome: Median Change in Asthma Score 2 Hours After Intervention
Description: The scale used is the Asthma Score published by Qureshi et al. The Asthma Score ranges from a low of 5 to maximum of 15 points. One to 3 points are given for each of 5 categories: age-based respiratory rate, oxygen saturation, wheeze, retractions, and dyspnea. For category detalails, please see the Qureshi reference. Scores of 5-7 are considered mild, 8-11 moderate, and 12-15 severe. Asthma Scores are recorded prior to any intervention and at 2 hours after budesonide inhalation suspension/albuterol intervention or saline placebo/albuterol comparator.
Time Frame: Initial asthma score minus score 2 hours after budesonide/albuterol intervention or saline placebo/albuterol comparator
Population: 88 of the 91 patients randomized to budesonide were evaluable for the primary outcome (1 was discharged home, 1 had no 2 hour score, and 1 did not have a valid initial score). 81 of the 89 patients randomized to placebo were evaluable (1 inadvertently received standard therapy, 2 withdrew, and 5 were admitted before a 2 hour score evaluation).
Measure: Median (Full Range); unit: Units on a scale
Arm/Group | Budesonide Inhalation Suspension (BIS) | Placebo (Normal Saline)
Number analyzed (Participants) | 88 | 81
Units on a scale | -3 [-8 to 2] | -3 [-8 to 3]
Statistical Analysis 1: Comparison: Budesonide Inhalation Suspension (BIS) vs Placebo (Normal Saline); Test type: Superiority or Other; p = 0.44, Wilcoxon (Mann-Whitney) — The difference in median improvement between treatment groups was expected to be greater than 2

2. Secondary Outcome: Number of Patients Hospitalized
Description: The number of patients requiring hospital admission 4 hours after budesonide/albuterol intervention or saline/albuterol comparator. All hospitalization decisions are made at the discretion of the attending physician.
Time Frame: within 4 hours after the budesonide/albuterol intervention or saline/albuterol placebo
Measure: Number; unit: Participants
Arm/Group | Budesonide Inhalation Suspension (BIS) | Placebo (Saline)
Number analyzed (Participants) | 91 | 89
Participants | 56 | 55
Statistical Analysis 1: Comparison: Budesonide Inhalation Suspension (BIS) vs Placebo (Saline); Test type: Superiority or Other; p = 0.97, Chi-squared; Risk Difference (RD) = 0.0, 95% CI 2-sided [-0.14 to 0.14]

3. Secondary Outcome: Change in Mean Heart Rate
Description: Mean of heart rate in beats per minute before treatment minus mean of heart rate 2 hours after treatment with either budesonide/albuterol or saline/albuterol
Time Frame: From the initial heart rate to heart rate 2 hours after intervention with budesonide/albuterol or saline/albuterol comparator
Measure: Mean (95% Confidence Interval); unit: Beats per minute
Arm/Group | Budesonide Inhalation Suspension (BIS) | Placebo (Normal Saline)
Number analyzed (Participants) | 82 | 72
Beats per minute | 12 [7 to 17] | 13 [9 to 17]
Statistical Analysis 1: Comparison: Budesonide Inhalation Suspension (BIS) vs Placebo (Normal Saline); Test type: Superiority or Other; t-test, 2 sided; Mean Difference (Net) = -1, 95% CI 2-sided [-7 to 6], Standard Error of Mean 3

4. Secondary Outcome: Mean Change in Respiratory Rate.
Description: Mean respiratory rate in breaths per minute before treatment minus respiratory rate 2 hours after treatment with either budesonide/albuterol or saline/albuterol comparator.
Time Frame: Initial rate, minus rate taken 2 hours after budesonide/albuterol intervention or saline/albuterol comparator
Measure: Mean (95% Confidence Interval); unit: Breaths per minute
Arm/Group | Budesonide Inhalation Suspension (BIS) | Placebo (Normal Saline)
Number analyzed (Participants) | 83 | 71
Breaths per minute | -6 [-8 to -3] | -6 [-8 to -4]
Statistical Analysis 1: Comparison: Budesonide Inhalation Suspension (BIS) vs Placebo (Normal Saline); Test type: Superiority or Other; t-test, 2 sided; Mean Difference (Net) = 0, 95% CI 2-sided [-3 to 3], Standard Error of Mean 1.6

5. Secondary Outcome: Oxygen Saturation.
Description: Mean oxygen saturation (non-invasive pulse-oximetry, % hemoglobin saturation) 2 hours after treatment with either budesonide/albuterol or saline/albuterol comparator minus mean oxygen saturation before treatment.
Time Frame: 2 hours after treatment with either budesonide/albuterol or saline/albuterol comparator
Measure: Mean (95% Confidence Interval); unit: Percent Hemoglobin Saturation
Arm/Group | Budesonide Inhalation Suspension (BIS) | Placebo (Normal Saline)
Number analyzed (Participants) | 72 | 64
Percent Hemoglobin Saturation | 1.0 [0.3 to 1.6] | 1.0 [0.2 to 1.7]
Statistical Analysis 1: Comparison: Budesonide Inhalation Suspension (BIS) vs Placebo (Normal Saline); Test type: Superiority or Other; t-test, 2 sided; Mean Difference (Net) = 0, 95% CI 2-sided [-1 to 1], Standard Error of Mean .49

6. Secondary Outcome: Number of Subjects Remaining in the Severe Asthma Category
Description: Of the patients who presented in the severe asthma category (Asthma Severity score of 12-15), those who remained in this category 2 hours after the budesonide/albuterol intervention or saline/albuterol comparator.
Time Frame: From the initial score to 2 hours after intervention with budesonide/albuterol or saline/albuterol comparator
Population: Number of patients who presented in the severe asthma category (Asthma Score 12-15) who remained in that category 2 hours after either the intervention with budesonide/albuterol or saline/albuterol comparator.
Measure: Number; unit: Participants
Arm/Group | Budesonide Inhalation Suspension (BIS) | Placebo (Normal Saline)
Number analyzed (Participants) | 35 | 27
Participants | 4 | 4
Statistical Analysis 1: Comparison: Budesonide Inhalation Suspension (BIS) vs Placebo (Normal Saline); Test type: Superiority or Other; p = 0.69, Chi-squared; Risk Difference (RD) = -0.03, 95% CI [-0.20 to 0.14]

7. Secondary Outcome: Number of Subjects Moving From the Severe Asthma to Moderate Asthma Category
Description: Of the patients who presented in the severe asthma category (Asthma Severity score of 12-15), those who moved to the moderate category (Asthma Severity score 8-11) 2 hours after the budesonide/albuterol intervention or saline/albuterol comparator.
Time Frame: From the initial score to 2 hours after intervention with budesonide/albuterol or saline/albuterol comparator
Population: Number of patients who presented in the severe asthma category (Asthma Score 12-15) who moved to the moderate asthma category (Asthma Score 8-11) 2 hours after either the intervention with budesonide/albuterol or saline/albuterol comparator.
Measure: Number; unit: Participants
Arm/Group | Budesonide Inhalation Suspension (BIS) | Placebo (Normal Saline)
Number analyzed (Participants) | 35 | 27
Participants | 22 | 11
Statistical Analysis 1: Comparison: Budesonide Inhalation Suspension (BIS) vs Placebo (Normal Saline); Test type: Superiority or Other; p = 0.08, Chi-squared; Risk Difference (RD) = 0.22, 95% CI 2-sided [-0.02 to 0.47]

8. Secondary Outcome: Number of Subjects Moving From the Severe Asthma to Mild Asthma Category
Description: Of the patients who presented in the severe asthma category (Asthma Severity score of 12-15), those who moved to the mild category (Asthma Severity score 5-7) 2 hours after the budesonide/albuterol intervention or saline/albuterol comparator.
Time Frame: From the initial score to 2 hours after intervention with budesonide/albuterol or saline/albuterol comparator
Population: as for outcome 7
Measure: Number; unit: Participants
Arm/Group | Budesonide Inhalation Suspension (BIS) | Placebo (Normal Saline)
Number analyzed (Participants) | 35 | 27
Participants | 8 | 10
Statistical Analysis 1: Comparison: Budesonide Inhalation Suspension (BIS) vs Placebo (Normal Saline); Test type: Superiority or Other; p = 0.22, Chi-squared; Risk Difference (RD) = -0.14, 95% CI 2-sided [-0.37 to 0.08]

9. Secondary Outcome: Relapse / Readmission Numbers.
Description: Participants admitted to the hospital within 5 days of the ED visit
Time Frame: within 5 days of ED visit
Population: 89 of the 91 patients randomized to BIS were available for follow-up. 85 of the 89 patients randomized to placebo were available.
Measure: Number; unit: Participants
Arm/Group | Budesonide Inhalation Suspension (BIS) | Placebo (Normal Saline)
Number analyzed (Participants) | 89 | 85
Participants | 2 | 2

10. Primary Outcome: Mean Change in Asthma Score at 2 Hours
Description: as for outcome 1
Time Frame: Initial asthma score minus score 2 hours after budesonide/albuterol intervention or saline placebo/albuterol comparator
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Budesonide Inhalation Suspension (BIS) | Placebo (Normal Saline)
Number analyzed (Participants) | 88 | 81
Units on a scale | -2.9 [-3.4 to -2.4] | -3.0 [-3.5 to -2.5]
Statistical Analysis 1: Comparison: Budesonide Inhalation Suspension (BIS) vs Placebo (Normal Saline); Test type: Superiority or Other; p = 0.78, t-test, 2 sided; Mean Difference (Net) = 0.1, 95% CI 2-sided [-0.6 to 0.8], Standard Error of Mean 0.36

11. Secondary Outcome: Number of Participants With Adverse Events (Non-serious).
Time Frame: within 30 days of the ED visit
Population: Of the 180 patients randomized, 91 were to BIS, 89 were to placebo. Two patients were lost to follow-up in the BIS group and 4 in the placebo group.
Measure: Number; unit: Participants
Arm/Group | Budesonide Inhalation Suspension (BIS) | Placebo (Normal Saline)
Number analyzed (Participants) | 89 | 85
Participants
  Rhinorrhea | 6 | 11
  Headache | 5 | 9
  Diarrhea | 3 | 7
  Sore throat | 4 | 3
  Cough | 2 | 3
  Hyperglycemia | 2 | 0

12. Secondary Outcome: Serious Adverse Events
Description: Serious Adverse Events
Time Frame: 0-5 days
Population: as for outcome 9
Measure: Number; unit: participants
Arm/Group | Budesonide Inhalation Suspension (BIS) | Placebo (Saline)
Number analyzed (Participants) | 89 | 85
participants
  Return within 5 days with hosptial admission | 2 | 2
  Increased level of care | 1 | 0

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Budesonide Inhalation Suspension (BIS) | Placebo (Saline)
Serious Adverse Events (participants affected / at risk) | 3/91 | 2/88
Other Adverse Events (participants affected / at risk) | 30/91 | 27/91
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Budesonide Inhalation Suspension (BIS) (N=91) | Placebo (Saline) (N=88)
Hospitalization within 5 days of Emergency Department discharge home (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Increased level of care (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Budesonide Inhalation Suspension (BIS) (N=91) | Placebo (Saline) (N=91)
rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 11 (11)
headache (Nervous system disorders) | 5 (5) | 9 (9)
diarrhea (Gastrointestinal disorders) | 3 (3) | 7 (7)
sore throat (Infections and infestations) | 4 (4) | 3 (3)
cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
hyperglycemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
emesis (Gastrointestinal disorders) | 4 (4) | 6 (6)
fever (Infections and infestations) | 3 (3) | 3 (3)
epistaxis (Blood and lymphatic system disorders) | 3 (3) | 1 (1)
ear infection (Infections and infestations) | 0 (0) | 3 (3)
respiratory infection (Infections and infestations) | 4 (4) | 1 (1)
stomach ache (Gastrointestinal disorders) | 1 (1) | 3 (3)
chest pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
leg pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No